CLINICAL TRIAL: NCT03746028
Title: The Lupus prEGnAnCY Cohort: An International Prospective Cohort of Lupus Pregnancies
Acronym: LEGACY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Duke University (Other); University of California, Los Angeles (Other); Dalhousie University (Other); Hanyang University (Other); Hospital for Special Surgery, New York (Other); Johns Hopkins University (Other); Monash University (Other); New York University (Other); Oklahoma Medical Research Foundation (Other); University of North Carolina (Other); Temple University (Other); University of Alabama at Birmingham (Other); University of Birmingham (Other); University of Calgary (Other); University of California (Other); University of Copenhagen (Other); University of Manitoba (Other); University of Michigan (Other); University of Toronto (Other); NYU Langone Health (Other); University of British Columbia (Other); National Institute of Medical Science & Nutrition (Unknown); Laval University (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Evelyne Vinet, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: LEGACY - MP-37-2018-3707 (MP); 384331 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2018-10-23; First posted 2018-11-19 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Systemic Lupus Erythematosus; Pregnancy Complications
Keywords: Adverse Pregnancy Outcomes; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — In order to achieve these objectives, clinical data and blood sample results obtained through the MUHC LEGACY Biobank (directed by Dr. Evelyne Vinet) will be analysed. The objective of the LEGACY Biobank (the "Bank") is the conservation of blood samples; more specifically, plasma, sera, and crude white cell pellet and clinical data ("material/data") collected from an international multi-centre prospective cohort of pregnant women with systemic lupus erythematosus (SLE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal is to evaluate adverse pregnancy outcomes (APO), their predictors and potential preventive therapies, such as aspirin (ASA). The investigator aims to improve the outcomes for women with SLE and offsprings. By quantifying the risk of APO conferred by clinical risk factors that can be assessed early in pregnancy (i.e. first trimester), health professionals could be better equipped to estimate the individual risk of SLE pregnancies and the need for heightened surveillance and guide counseling for prophylactic measures, including ASA. Moreover findings from this study could eventually lead to the choice and weighting of first trimester clinical factors in future clinical prediction models for APO in SLE. The investigator's research efforts will improve reproductive health of SLE women, "mitigating the damage, functional loss, and disability that result from a chronic inflammatory disorder", such as SLE.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) predominantly affects women during their reproductive years. As SLE is associated with substantial fetal and maternal morbidity during pregnancy and beyond it is crucial to identify predictors of adverse pregnancy outcomes (APO) in SLE to appropriately counsel patients and guide monitoring during pregnancy. SLE pregnancies result in high rates of preterm birth, preeclampsia and fetal loss compared to pregnancies in unaffected women.

As a prior effort to address this issue, team members performed a large prospective study (the PROMISSE study) to determine baseline predictors of APO in SLE women with inactive and mild/moderate disease activity. However, PROMISSE included a selected population, which might not be representative of all SLE women particularly those with severe disease activity and/or active nephritis. Furthermore new data suggest that antiphosphatidylserine/prothrombin antibodies (aPS/PT), which are antiphospholipid antibodies (aPL), are strongly associated with APO. These antibodies were not evaluated in the PROMISSE study, or any other study of SLE pregnancies to date. Moreover, despite evidence of the beneficial effect of aspirin (ASA) in non-SLE women at high risk of APO, there are currently no studies of ASA in SLE pregnancies. This is a critical knowledge gap as ASA could have a large benefit for SLE mothers and their offspring.

The goal is to evaluate adverse pregnancy outcomes (APO), their predictors, and potential preventive therapies. The investigator aims to improve the outcomes for women with SLE and their offspring. Primary outcomes of this study are to determine the risk of APO in this cohort, as well as to evaluate the patterns of ASA use in the LEGACY cohort. Secondary outcomes will be to conduct pilot analyses to assess baseline predictors of APO determined in the PROMISSE study (i.e. lupus anticoagulant (LAC) positivity, antihypertensive use, platelets level, race/ethnicity, prior nephritis, disease activity), and to evaluate prevalence of aPS/PT in SLE pregnancies.

Design: In order to achieve these objectives, clinical data and blood sample results obtained through the McGill University Health Centre (MUHC) LEGACY Biobank (directed by Dr. Evelyne Vinet) will be analyzed. Patient recruitment, consent, management and storage of data/samples will be done in accordance with the Biobank Management Framework. The LEGACY Biobank informed consent forms will be used to obtain participant consent.

Methodology: Research activities will be conducted in accordance with the LEGACY Biobank Management Framework. English and French speaking pregnant SLE women will be enrolled up to and including the 16 6/7 weeks regardless of disease manifestations, level of disease activity and drug exposures. Pregnancies up to and including 12 weeks gestation will be targeted but pregnancies up until 16 6/7 weeks will be included. The attending staff or a nurse not involved with the study or the administrative assistant will introduce the study to pregnant women with Lupus. If patients are interested in learning more patients will be approached by coordinator who will explain the study in detail.

The main outcome of interest will be APO, which will be defined (as in PROMISSE) as a composite of specific outcomes including either: 1) fetal death after 20 weeks gestation, 2) neonatal death due to preterm birth and/or placental insufficiency 3) preterm delivery or termination of pregnancy <36 weeks due to placental insufficiency, gestational hypertension, preeclampsia and/or eclampsia and/or 4) small for gestational age neonate (i.e. birth weight <5th percentile).

Patients will be reassessed in the 2nd and 3rd trimesters and postpartum (8-12 weeks after delivery). The investigator will calculate the risk of APO as a function of gestational age, with the Kaplan-Meier estimator. The investigator will use descriptive statistics to measure the prevalence of ASA use at baseline and compare the prevalence of use across all trimesters. Exploratory analyses will examine correlates of ASA initiation and non-adherence during pregnancy, using univariate regression analyses, evaluating relevant baseline covariates. The investigator will calculate descriptive statistics to assess and compare the baseline prevalence of positive aPS/PT and LAC in SLE pregnancies with and without APO. In pilot univariate analyses, the investigator will evaluate if baseline covariates as determined in the PROMISSE study (i.e. LAC, antihypertensives, platelets, race/ethnicity, nephritis, disease activity) correlate with APO.

Confidentiality: All data/samples used in this project will be obtained from the MUHC research ethics board (REB) approved LEGACY Biobank. Patient recruitment and informed consent will be obtained as per the procedures described in the management framework. This study will be conducted in accord with Tri-Council Policy Statement.

Collection of socio-demographic, clinical data and reasons for refusal will be conserved anonymously from patients refusing to participate in the bank. This information will be included in the statistical analysis in order to assess selection bias, that is, if patients who refuse participation may be a little different (in terms of age, sex, socioeconomic status, etc) from those who do participate.Only data relevant to this study will be collected by the research team from the bank. All the information collected during the research project will remain confidential to the extent required and provided by law.

Statistical Analysis:

Estimating the Risk of APO (Primary Objective 1): The investigator will calculate the risk of APO as a function of gestational age, with the Kaplan-Meier estimator. By using gestational age as the time axis, the investigator appropriately uses a cohort of conceptions rather than a cohort of births as the study sample for fetal complications. This approach is referred to as the "fetus-at-risk" approach.

Pattern of ASA Use (Primary Objective 2): The investigator will use descriptive statistics to measure the prevalence of ASA use at baseline and compare the prevalence of use across all trimesters. In addition the investigator will determine the proportion of patients who initiated ASA during pregnancy and the proportion of subjects already on ASA prior to pregnancy, exploring indications of use. The investigator will measure the frequencies of dosage used (i.e. 80 mg, 160 mg, and 325 mg). Exploratory analyses will examine correlates of ASA initiation and ASA non-adherence, during pregnancy using a univariate regression analysis estimated with the generalized estimating equation (GEE) method, evaluating the following baseline covariates: maternal age, race/ethnicity, obesity, aPL autoantibodies, prior preeclampsia, prior nephritis, and anti-hypertensive use.

Estimates for Predictors of APO (Secondary Objectives): The investigator will perform pilot univariate Cox proportional hazards regression analyses with frailties, using gestational age as the time axis. As mentioned this approach called the "fetus-at-risk" approach refers to the use of cohorts of conceptions (by using gestational age as the time axis) rather than cohorts of births, as the appropriate study sample for fetal complications. In these pilot univariate analyses, investigator will evaluate if baseline covariates as determined in the PROMISSE study (i.e. LAC positivity, antihypertensive use, platelets level, race/ethnicity, prior nephritis, disease activity as measured by the PGA) predict APO, exploring additional risk factors such as nulliparity, maternal age, pre-gestational diabetes, obesity (BMI above 30) and medication use (corticosteroids, antimalarials, immunosuppressive and low-dose aspirin).

aPS/PT Prevalence (Secondary Objectives): The investigator will calculate descriptive statistics to assess and compare the prevalence at baseline of positive aPS/PT and LAC in SLE pregnancies with and without APO. In pilot analyses, the investigator will perform a univariate Cox proportional hazards regression analysis with frailties to explore if aPS/PT predict APO. These secondary analyses are not meant to be definitive but rather allow the investigator to make precise power calculations for a more definitive trial funded by future applications.

Timeline: In the first 10 months patient recruitment and follow up will occur with concurrent data entry. In the following month the investigator will perform analyses assessing the risk of APO and the pattern of ASA use in ongoing and completed pregnancies. The investigator will also conduct pilot analyses to determine the baseline prevalence of aPS/PT in pregnant SLE women comparing those with and without APO. In last month the investigator will finalize interpretation of results and prepare results for presentation at national and international scientific meetings and complete at least 3 manuscripts for publication in a peer review journal.

Dissemination of Results: The measurement of success will go beyond the timely completion of each objective, the publications anticipated from the investigator's research and the successful application to additional funding opportunities. The project will offer a unique opportunity of integrated knowledge translation (KT). The investigator will disseminate the data generated by the proposal at different levels (public, patients, government etc) through various venues (meetings, websites, publications etc). The investigator plans to hold one stakeholder workshop and engage with key stakeholders including patient advocacy groups such as Lupus Canada and Lupus Foundation of America and representatives of public health agencies. The investigator has a proven track record in this area. Dr Vinet is leading the subgroup dealing with reproductive issues in development of Canadian recommendations on the monitoring and care of patients with SLE. The findings will help inform these efforts.

Possible Limitations: A possible limitation to the study is the lack of harmonization in the collection of samples/data. The team of investigators has a very long history (over decades) of working together in national (Canadian Network for Improved Outcomes in SLE, CaNIOS) and international (SLICC) groups. These research networks have established methods for standardized sample and data collection. However ongoing compliance of this standardization will be monitored to ensure that efforts will indeed yield results that are generalizable across SLE populations. The investigator will review sample and data collection protocols with investigators and coordinators offering monthly teleconferences and summaries of recruitment and data collection as feedback for investigators.

Loss to follow-up is always a potential problem but in general loss to follow-up in SLE cohorts is low (due to the fact that patients are not only being studied but are receiving care) and in a pregnancy cohort, follow up is often very high, as pregnancy is a time when women are particularly inclined to be adherent to visits. In PROMISSE, loss to follow-up was very rare, occurring in less than 1% of subjects.

Expected Outcomes: The investigator hypothesizes that APO rates will be higher in the LEGACY cohort (an unselected cohort of SLE pregnancies) versus the PROMISSE cohort. In addition despite the increased risk of APO, the investigator hypothesizes that at least one third of SLE pregnancies will not be exposed to ASA before 16 weeks of gestation. The investigator expects that the prevalence of aPS/PT in SLE pregnancies with APO will be higher than in SLE pregnancies without APO.

ELIGIBILITY:
Patient recruitment, consent, management and storage of data/samples will be done in accordance with the Biobank Management Framework. The LEGACY Biobank informed consent forms will be used to obtain participant consent.

Inclusion criteria:

1. Pregnant women with a SLE diagnosis based on the SLICC classification criteria;
2. Followed at participating sites;
3. English and French speaking;
4. Gestational age up to 16-6/7 weeks* inclusively
5. Between the ages of 18 and 45 years;
6. More than one pregnancy per subject is allowed for the LEGACY Biobank; however, only one pregnancy per subject will be included for women taking part in the Aspirin patterns of use and adherence for preeclampsia in SLE pregnancies;
7. Single and multiple intrauterine pregnancies are permitted. *Our aim is to recruit subjects under or equal to 12 weeks but we will include pregnancies up to 16-6/7 weeks inclusively.

Exclusion Criteria

1. Pregnant women who do not meet the SLE diagnosis based on the SLICC classification;
2. Women who are not followed at participating sites;
3. Women who do not speak English or French;
4. Gestational age at 17 weeks and above;
5. Under the age of 18 and over the age of 45;
6. Men are not eligible for this biobank;
7. Women with extrauterine pregnancies;
8. Women who cannot provide informed consent due to severe illness;
9. Women who are cognitively impaired or incapable of understanding the text written on the consent form.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: In accordance with the Biobank Management Framework. Participation will take place at the Systemic Lupus International Collaborating Clinics (SLICC) centres in Canada (including the Montreal General Hospital), in the United States, and in Mexico, Denmark, South Korea, and Australia. (The SLICC group represents rheumatologists interested in lupus from over 30 centres and 14 countries with a strong publication record in lupus research.) Recruitment will also take place at other sites that are not part of the SLICC group in Canada and the United States.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Risk of adverse pregnancy outcomes in pregnant women with SLE | Up until 28 days after end of pregnancy
  Fetal death, neonatal death, preterm delivery or termination of pregnancy, and small for gestational age neonate confirmed by chart review and autopsy report.
Change in patterns of ASA use in the LEGACY cohort from baseline ( <or equal to 12 weeks gestation) to end of pregnancy | From ≤ 12 weeks gestation (baseline) to 8-12 weeks after delivery (postpartum)
  The Adherence to Refills and Medications Scale (ARMS), a validated self-reported questionnaire developed for patients with chronic disease with low literacy, measures ASA adherence. A self-reported aspirin adherence questionnaire consisting of 3 to 6 questions about the use of aspirin during current pregnancy measures ASA use. A visual analogue scale from 0 to 10 measures frequency of ASA ingestion. Change in ASA use will be measured by the questionnaires. Frequencies of dosage of ASA will also be measured.

SECONDARY OUTCOMES:
Baseline predictors of adverse pregnancy outcomes | First trimester (up to 20 weeks)
  Baseline covariates such as lupus anticoagulant antibodies, a subtype of anticoagulant antibodies, Antiphosphatidylserine/prothrombin antibodies (aPS/PT), antihypertensive use, disease activity, platelet levels will be measured and defined by the physician-in-charge. Nephritis history, race/ethnicity, nulliparity, maternal age, pre-gestational diabetes, obsesity (BMI above 30) and medication use (corticosteroids, antimalarials, immunosuppressive and low-dose aspirin) will be characterized.
  Measures for disease activity include the SLE Pregnancy Disease Activity Index (SLEPDAI), a widely-recognized adaptation of the validated SLE Disease Activity Index, reflects disease activity in pregnancy context.
Comparison of Antiphosphatidylserine/prothrombin antibodies (aPS/PT) in SLE pregnancies from ≤ 12 weeks pregnant (baseline) to 8-12 weeks after delivery (postpartum) | From ≤ 12 weeks gestation (baseline) to 8-12 weeks after delivery (postpartum)
  Positive results for Antiphosphatidylserine/prothrombin antibodies (aPS/PT) and and lupus anticoagulant results in pregnant women with SLE with and without adverse pregnancy outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Vinet, MD/PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Information will be kept between investigators.

REFERENCES:
- [Background] Buyon JP, Kim MY, Guerra MM, Laskin CA, Petri M, Lockshin MD, Sammaritano L, Branch DW, Porter TF, Sawitzke A, Merrill JT, Stephenson MD, Cohn E, Garabet L, Salmon JE. Predictors of Pregnancy Outcomes in Patients With Lupus: A Cohort Study. Ann Intern Med. 2015 Aug 4;163(3):153-63. doi: 10.7326/M14-2235. PMID 26098843
- [Background] Petri M, Allbritton J. Fetal outcome of lupus pregnancy: a retrospective case-control study of the Hopkins Lupus Cohort. J Rheumatol. 1993 Apr;20(4):650-6. PMID 8496859
- [Background] Georgiou PE, Politi EN, Katsimbri P, Sakka V, Drosos AA. Outcome of lupus pregnancy: a controlled study. Rheumatology (Oxford). 2000 Sep;39(9):1014-9. doi: 10.1093/rheumatology/39.9.1014. PMID 10986308
- [Background] Clowse ME, Jamison M, Myers E, James AH. A national study of the complications of lupus in pregnancy. Am J Obstet Gynecol. 2008 Aug;199(2):127.e1-6. doi: 10.1016/j.ajog.2008.03.012. Epub 2008 May 5. PMID 18456233
- [Background] Al Arfaj AS, Khalil N. Pregnancy outcome in 396 pregnancies in patients with SLE in Saudi Arabia. Lupus. 2010 Dec;19(14):1665-73. doi: 10.1177/0961203310378669. Epub 2010 Oct 14. PMID 20947541
- [Background] Ko HS, Ahn HY, Jang DG, Choi SK, Park YG, Park IY, Lee G, Park SH, Shin JC. Pregnancy outcomes and appropriate timing of pregnancy in 183 pregnancies in Korean patients with SLE. Int J Med Sci. 2011;8(7):577-83. doi: 10.7150/ijms.8.577. Epub 2011 Oct 1. PMID 22022210
- [Background] Liu J, Zhao Y, Song Y, Zhang W, Bian X, Yang J, Liu D, Zeng X, Zhang F. Pregnancy in women with systemic lupus erythematosus: a retrospective study of 111 pregnancies in Chinese women. J Matern Fetal Neonatal Med. 2012 Mar;25(3):261-6. doi: 10.3109/14767058.2011.572310. Epub 2011 Apr 19. PMID 21504337
- [Background] Shand AW, Algert CS, March L, Roberts CL. Second pregnancy outcomes for women with systemic lupus erythematosus. Ann Rheum Dis. 2013 Apr;72(4):547-51. doi: 10.1136/annrheumdis-2011-201210. Epub 2012 Jun 29. PMID 22753385
- [Background] Smyth A, Oliveira GH, Lahr BD, Bailey KR, Norby SM, Garovic VD. A systematic review and meta-analysis of pregnancy outcomes in patients with systemic lupus erythematosus and lupus nephritis. Clin J Am Soc Nephrol. 2010 Nov;5(11):2060-8. doi: 10.2215/CJN.00240110. Epub 2010 Aug 5. PMID 20688887
- [Background] Joseph KS. The fetuses-at-risk approach: clarification of semantic and conceptual misapprehension. BMC Pregnancy Childbirth. 2008 Mar 26;8:11. doi: 10.1186/1471-2393-8-11. PMID 18366767
- See also: James G, Witten D, Hastie T, Tibshirani R. An Introduction to Statistical Learning-With Applications in R. New York: Springer; 2013. — http://www.springer.com/gp/book/9781461471370